CLINICAL TRIAL: NCT02207738
Title: Comparative Study of Efficacy and Safety Between Fractional Microneedling Radiofrequency and Bipolar Radiofrequency Treatment for Acne Scar
Brief Title: Comparison of Efficacy Between Fractional Microneedling Radiofrequency and Bipolar Radiofrequency for Acne Scar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-1062
Record Dates: First submitted 2014-06-26; First posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Acne; Scar
Keywords: acne; acne scar; microneedling radiofrequency; bipolar radiofrequency
MeSH Terms: conditions — Acne Vulgaris; Cicatrix

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- microneedling radiofrequency device (Experimental): microneedling radiofrequency
  Interventions: Device: microneedling radiofrequency device
- bipolar radiofrequency device (Active Comparator): bipolar radiofrequency treatment
  Interventions: Device: bipolar radiofrequency

INTERVENTIONS:
Device: microneedling radiofrequency device — Microneedling radiofrequency device is composed of 49 insulated microneedle which emit radiofrequency from the needle tip. This radiofreqeuncy generates dermal heat which evokes biological effect.
  Other Names: INFINI(Lutronics, Goyang, Korea)
  Arms: microneedling radiofrequency device
Device: bipolar radiofrequency — bipolar radiofrequency instrument gives out bipolar radiofrequency from the hand piece tip. This bipolar radiofrequency generates dermal heat which has a lot of bilogical effect.
  Other Names: Polaris(syneron, israel)
  Arms: bipolar radiofrequency device

SUMMARY:
Compare the efficacy and safety profile of microneedling radiofrequency and that of bipolar radiofrequency treatment for acne scar.

DETAILED DESCRIPTION:
Efficacy and safety of microneedling radiofrequency for acne scar Efficacy and safety bipolar radiofrequency treatment for acne scar compare the efficacy and safety profile of microneedling radiofrequency and that of bipolar radiofrequency treatment for acne scar

ELIGIBILITY:
Inclusion Criteria:

* moderate acne scar
* mild to moderate acne lesions

Exclusion Criteria:

* taking acne medication oral drugs within 2 months topical drugs within 2 weeks
* taken anu procedures for acne scar within 6 months
* taking steroid,nonsteroidal antiinflammtory drugs, isotretinoin
* underlying diabetes mellitus, keloid, or any malignancy

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Global assessment of acne scar | 12 weeks
  5-point grading of acne scar quartile assessment of acne scar improvement through comparing the photos taken before treatment and after treatment

SECONDARY OUTCOMES:
ECCA | 12 weeks
  quantitative assessment of acne scar ECCA assessment is established by previous article. this method quantifies severity of acne scar by counting the number of acne scar categorized by their shape. Then, the number of scars are multiplied by weighing factors determined by scar types. ECCA is the total sum of these points. please refer the Dreno et al, Dermatology, 2007;214:46-51
Adverse effect | 12 weeks
  adverse effects were measured by Epithelization Scale. ES is the total sum of evaluation of three components after wounding. please refer this article Min et al, Wound Repair and Regen, 2014;22(2):212-9

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hun Suh, PhD, Study Chair — Department of Dermatology, Seoul National University College of Medicine; Seonguk Min, Msc, Principal Investigator — Department of Dermatology, Seoul National University College of Medicine
Locations (1):
- Department of Dermatology, Seoul National University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Yeung CK, Chan NP, Shek SY, Chan HH. Evaluation of combined fractional radiofrequency and fractional laser treatment for acne scars in Asians. Lasers Surg Med. 2012 Oct;44(8):622-30. doi: 10.1002/lsm.22063. Epub 2012 Aug 16. PMID 22899398